CLINICAL TRIAL: NCT01618461
Title: PictureRx: An Intervention to Reduce Latino Health Disparities (Supplement: Medical Icons)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PictureRx, LLC (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, M Brian Riley, Director of Research, PictureRx, LLC
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 3R43MD004048-02S1 (NIH); 3R43MD004048-02S1 (NIH)
Record Dates: First submitted 2012-06-11; First posted 2012-06-13 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Understanding of Medication Instructions; Recall of Medication Instructions
Keywords: Prescription drug information; Medication management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Text instructions (No Intervention): Medication instructions displayed in text format
- Drug indication icons (Experimental): Icons illustrate the purpose of each medication
  Interventions: Behavioral: Drug indication icons
- Structured instructions (Experimental): Graphical format shows what time(s) of day each medication should be taken
  Interventions: Behavioral: Structured instructions
- Icons + Structured instructions (Experimental): Icons illustrate the purpose of each medication, and a graphical format shows what time(s) of day each medication should be taken
  Interventions: Behavioral: Drug indication icons; Behavioral: Structured instructions

INTERVENTIONS:
Behavioral: Drug indication icons — Icons illustrate the purpose of each medication
  Arms: Drug indication icons; Icons + Structured instructions
Behavioral: Structured instructions — Graphical format shows what time(s) of day each medication should be taken
  Arms: Icons + Structured instructions; Structured instructions

SUMMARY:
Research shows that well-developed icons and other pictorials aid in the comprehension of medication information and are effective in improving patients' medication management. This experimental study seeks to test the effect of icons and structured medication information on subjects' processing and recall of simulated medication instructions in a computer testing environment. The study planned to enroll 200 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years old
* Fluency in English or Spanish
* Manage their own prescription medicines, and
* Be taking at least one chronic medication

Exclusion Criteria:

* Too ill to complete the experiment
* Having visual acuity worse than 20/50 via Rosenbaum Visual Acuity exam (eyechart)
* Inability to communicate in either Spanish or English
* Overt psychiatric illnesses, overt delirium or dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Understanding of medication instructions | Within 10-20 minutes
  Participants' ability to state the drug indication

SECONDARY OUTCOMES:
Recall of medication instructions | Within 10-20 minutes
  Participants' ability to recall the instructions after viewing a series of medications

CONTACTS AND LOCATIONS:
Overall Officials: M Brian Riley, MA, Principal Investigator — PictureRx, LLC
Locations (2):
- United States (2):
  - Saint Thomas Family Health Center - West, Nashville, Tennessee
  - Saint Thomas Family Health Center - South, Nashville, Tennessee